CLINICAL TRIAL: NCT04846205
Title: Assessment of the Relationship Between Sleep Apnea Syndrome and Patent Foramen Ovale Among Young Subjects Victims of Cryptogenic Ischemic Stroke
Brief Title: Relationship Between Sleep Apnea Syndrome and Patent Foramen Ovale Among Victims of Cryptogenic Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN212021/CHUSTE
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Apnea Syndrome; Stroke
Keywords: obstructive sleep apnea syndrome; permeable foramen oval
MeSH Terms: conditions — Sleep Apnea Syndromes; Stroke; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent a systematic etiological: Patients who underwent a systematic etiological assessment in the context of their cryptogenic ischemic stroke between 2015 and 2020. A collect data in medical record will be realized.
  Interventions: Diagnostic Test: systematic etiological

INTERVENTIONS:
Diagnostic Test: systematic etiological — Theses following tests are made as usual practice :
  * Ventilator polygraphy, or polysomnography between 1 month and 1 year after cryptogenic ischemic stroke.
  * Transoesophageal ultrasound

SUMMARY:
Obstructive sleep apnea syndrome (OSAS) and patent foramen ovale (FOP) are considered as risk factors for stroke. OSAS generates a pressure increase in the right cavity during inspiratory efforts, which increases the number of right-left shunt embolus and therefore the risk of stroke. OSA and FOP are often thought as two separate entities, however, due to their high frequencies, they sometimes coexist and can influence the pathophysiology of each other. More researches are needed in this area to confirm this complex association and its role in triggering stroke.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) and patent foramen ovale (PFO) are considered as risk factors for stroke. In most cases, the presence of FOP has no clinical impact. Certain hemodynamic conditions inducing a right-left pressure gradient can promote the reopening of a FOP and allow the passage of blood, presenting micro or macro-thrombi, from the venous system to the arterial system, explaining the mechanism of paradoxical embolism. OSAS generates a pressure increase in the right cavity during inspiratory efforts, which increases the number of right-left shunt embolus and therefore the risk of stroke. OSA and FOP are often thought as two separate entities, however, due to their high frequencies, they sometimes coexist and can influence the pathophysiology of each other. Evidence of a clinically significant interaction and causation in the genesis of stroke remains limited. More researches are needed in this area to confirm this complex association and its role in triggering stroke.

ELIGIBILITY:
Inclusion Criteria:

- Patients who have had a cerebral or retinal infarction confirmed by brain imaging or a defined transient ischemic attack without an identifiable cause after a detailed etiological assessment

Exclusion Criteria:

* Identification of a cause of ischemic stroke:

  * Atheromatous stenosis > 50% (or atherosclerotic plaque < 50% threatening) of supra aortic trunk or intracranial arteries on echodoppler of the supra aortic trunk and transcranial or scanner angiography.
  * Emboligenic heart disease : atrial fibrillation and atrial flutter, thrombus in left atrium, spontaneous contrast in left atrium, decreased atrial flow, left ventricular ejection fraction (LVEF) < 40%, LV aneurysma, left intraventricular thrombus, recent myocardial infarction, cardiomyopathy ventricular dilated left with LVEF < 35%, mitral stenosis, prosthetic mitral or aortic valve, infectious and non-infectious endocarditis, valve or mural tumor, complicated aortic arch atheroma (plaque > = 4 mm, ulcerated plaque, thrombus on plaque), aortic dissection
  * Lacunar infarction symptomatic = < 1.5 cm on the CT scan, = < 2 cm on the diffusion MRI or the FLAIR.
  * No atherosclerotic arteriopathy : dissection, primary and secondary angitis, spastic angiopathy, etc…
  * Coagulopathy to come a long-term anticoagulant treatment (> 6 months) (anti-phospholipid syndrome, thrombophilia).
  * Blood disorders and cancer
  * Recent intravenous drug use (in the 6 months before the stroke).
  * Other potential causes:
* Severe respiratory impairment or pulmonary arterial hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who underwent a systematic etiological assessment in the context of their cryptogenic ischemic stroke between 2015 and 2020.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index | 1 year after the ischemic stoke
  Apnea Hypopnea Index (AHI) > 15 / h on ventilator polygraphy (PV), or AHI >10/h on polysomnography (PSG) will be considered as a risk factor

SECONDARY OUTCOMES:
Presence of foramen oval | 1 year after the ischemic stoke
  Presence of a foramen oval on transoesophageal ultrasound during the etiological assessment of the stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe CAMDESSANCHE, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No